CLINICAL TRIAL: NCT00295009
Title: A Multi-Center, Prospective, Randomized, Controlled Clinical Trial Comparing the Safety and Effectiveness of ProDisc to Spinal Fusion Surgery in the Treatment of Discogenic Pain Associated With DDD in the Lumbosacral Spine
Brief Title: Safety and Effectiveness Study of Prodisc to Spinal Fusion Surgery
Acronym: PDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDL-07272001
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases | interventions — Spinal Fusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1-Level Fusion (Active Comparator): Spinal fusion at a single lumbar level.
  Interventions: Procedure: Spinal Fusion
- 1-Level ProDisc (Experimental): Total disc replacement with the ProDisc device at one spinal lumbar level.
  Interventions: Device: ProDisc
- 2-Level Fusion (Active Comparator): Spinal fusion at two adjacent lumbar levels.
  Interventions: Procedure: Spinal Fusion
- 2-Level ProDisc (Experimental): Total disc replacement with the ProDisc device at two adjacent lumbar levels.
  Interventions: Device: ProDisc
- 1-level ProDisc (non-randomized) (Experimental): Total disc replacement with the ProDisc device for non-randomized subjects at one spinal lumbar level.
  Interventions: Device: ProDisc
- 2-Level ProDisc (Continued Access) (Active Comparator): Total disc replacement with the ProDisc device for non-randomized subjects at two spinal lumbar levels (only followed out to 24 months)
  Interventions: Device: ProDisc

INTERVENTIONS:
Device: ProDisc — Total disc replacement with ProDisc
  Arms: 1-Level ProDisc; 1-level ProDisc (non-randomized); 2-Level ProDisc; 2-Level ProDisc (Continued Access)
Procedure: Spinal Fusion — A circumferential fusion will be utilized as the control group in this study. The technique will consist of an interbody fusion procedure using commercially available femoral ring allograft. A posterior lateral fusion with autogenous iliac crest bone graft, combined with pedicle screw instrumentation.
  Arms: 1-Level Fusion; 2-Level Fusion

SUMMARY:
The objective of this clinical investigation is to compare the safety and effectiveness of ProDisc total disc replacement to spinal fusion surgery in the treatment of discogenic pain associated with DDD in the lumbosacral spine. There will be separate study arms for one and two level cases.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative Disc Disease (DDD) in one or two adjacent vertebral levels between L3 and S1. Diagnosis of DDD requires: a)Back and/or leg (radicular) pain; and b)Radiographic confirmation of any 1 of the following by CT, MRI, discography, plain film, myelography and/or flexion/extension films: Instability (greater than or equal to 3mm translation or 5° angulation); Decreased disc height >2mm; Scarring/thickening of annulus fibrosis; Herniated nucleus pulposus; or Vacuum phenomenon.
* Age between 18 and 60 years.
* Failed at least 6 months of conservative treatment.
* Oswestry Low Back Pain Disability Questionnaire score of at least 20/50 (40%)(Interpreted as moderate/severe disability).
* Psychosocially, mentally and physically able to fully comply with this protocol including adhering to follow-up schedule and requirements and filling out forms.
* Signed informed consent.

Exclusion Criteria:

* No more than 2 vertebral levels may have DDD and all diseased levels, either one or two, must be treated.
* Patients with involved vertebral endplates dimensionally smaller than 34.5mm in the medial-lateral and/or 27mm in the anterior-posterior directions.
* Known allergy to titanium, polyethylene, cobalt, chromium, or molybdenum.
* Prior fusion surgery at any vertebral level.
* Clinically compromised vertebral bodies at the affected level(s) due to current or past trauma.
* Radiographic confirmation of facet joint disease or degeneration.
* Lytic spondylolisthesis or spinal stenosis.
* Degenerative spondylolisthesis of grade >1.
* Back or leg pain of unknown etiology.
* Osteopenia or Osteoporosis: A screening questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen patients to determine if a DEXA scan is required. If DEXA is required, exclusion will be defined as a DEXA bone density measured T score less than
* 1.0. The World Health Organization defines osteoporosis as a DEXA T score less than or equal to -2.5.
* Paget's disease, osteomalacia or any other metabolic bone disease (excluding osteoporosis which is addressed above).
* Morbid obesity defined as a body mass index >40 or a weight more than 100 lbs. over ideal body weight.
* Pregnant or interested in becoming pregnant in the next 3 years.
* Active infection - systemic or local.
* Taking medication or any drug known to potentially interfere with bone/soft tissue healing (e.g., steroids).
* Rheumatoid arthritis or other autoimmune disease.
* Systemic disease including AIDS, HIV, Hepatitis.
* Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there has been no clinical signs or symptoms of the malignancy for at least 5 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 852 (Actual)
Dates: Start 2001-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

REFERENCES:
- [Derived] Zigler JE, Glenn J, Delamarter RB. Five-year adjacent-level degenerative changes in patients with single-level disease treated using lumbar total disc replacement with ProDisc-L versus circumferential fusion. J Neurosurg Spine. 2012 Dec;17(6):504-11. doi: 10.3171/2012.9.SPINE11717. Epub 2012 Oct 19. PMID 23082849

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-Level Fusion: Circumferential fusion at a single lumbar level.
- 1-Level ProDisc: Total disc arthroplasty with the ProDisc device at one spinal lumbar level.
- 1-Level ProDisc (Non-Randomized): Non-randomized total disc arthroplasty with the ProDisc device at one spinal lumbar level.
- 2-Level Fusion: Circumferential fusion at two adjacent lumbar levels.
- 2-Level ProDisc: Total disc arthroplasty with the ProDisc device at two adjacent lumbar levels.
- 2-Level ProDisc (Continued Access): Non-randomized total disc arthroplasty with the ProDisc device at two spinal lumbar levels. Continued Access patients only followed out to 24 months.
Period: Overall Study
Arm/Group | 1-Level Fusion | 1-Level ProDisc | 1-Level ProDisc (Non-Randomized) | 2-Level Fusion | 2-Level ProDisc | 2-Level ProDisc (Continued Access)
Started | 93 | 183 | 51 | 82 | 174 | 269
Treated | 80 | 162 | 50 | 72 | 165 | 259
Completed 24 Month Analysis | 71 | 148 | 45 | 60 | 133 | 198
Completed | 52 (Completed 60 month visit) | 134 (Completed 60 month visit) | 39 (Completed 60 month visit) | 57 (Completed 60 month visit) | 116 (Completed 60 month visit) | 0 (Continued Access patients were only followed out to 24 months)
Not Completed | 41 | 49 | 12 | 25 | 58 | 269

BASELINE CHARACTERISTICS:
Population: Enrolled and treated
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Level Fusion | 1-Level ProDisc | 1-Level ProDisc (Non-randomized) | 2-Level Fusion | 2-Level ProDisc | 2-Level ProDisc (Continued Access) | Total
Number analyzed (Participants) | 80 | 162 | 50 | 72 | 165 | 259 | 788
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (7.6) | 39.6 (8.0) | 37.9 (8.0) | 41.8 (7.8) | 41.8 (7.7) | 40.5 (7.4) | 40.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 79 | 30 | 33 | 70 | 103 | 358
  Male | 37 | 83 | 20 | 39 | 95 | 156 | 430
Region of Enrollment [Number; unit: participants]
  United States | 80 | 162 | 50 | 72 | 165 | 259 | 788

OUTCOME MEASURES:

1. Primary Outcome: Overall Success
Description: Overall success was a composite endpoint.
  A ProDisc patient was considered an overall success if, and only if, ALL of the following criteria were met:
  1. ODI score improved by at least 15% from baseline;
  2. SF-36 score improved from baseline;
  3. Neurologic parameters maintained or improved from baseline;
  4. No re-operations to modify or remove the implant; and
  5. Independent radiographic review confirmed no migration/subsidence, radiolucency, loss of disc height, loss of range of motion, or boney fusion.
  A Fusion patient was a considered to be a success if, and only if, ALL of the following criteria were met:
  1. Same as above
  2. Same as above
  3. Same as above
  4. No re-operations to modify the fusion site or correct a complication with an implant; and
  5. Independent radiographic review confirmed strong evidence of fusion and no motion, visible gaps in fusion mass, loss of disc height, migration/subsidence, implant loosening, halos, or radiolucencies
Time Frame: 24 Months
Population: Patients who completed all 24 month visit analyses
Measure: Number; unit: percentage of overall successes
Arm/Group | 1-Level Fusion | 1-Level ProDisc | 1-Level ProDisc (Non-randomized) | 2-Level Fusion | 2-Level ProDisc | 2-Level ProDisc (Continued Access)
Number analyzed (Participants) | 71 | 148 | 45 | 60 | 133 | 198
percentage of overall successes | 45.1 | 63.5 | 66.7 | 53.3 | 59.4 | 58.6

2. Primary Outcome: Overall Success
Description: Overall success was a composite endpoint. A ProDisc patient was considered an overall success if, and only if, ALL of the following criteria were met:
  1. ODI score improved by at least 15% from baseline;
  2. SF-36 score improved from baseline;
  3. Neurologic parameters maintained or improved from baseline;
  4. No re-operations required to modify or remove the implant; and
  5. Independent radiographic review confirmed no migration/subsidence, radiolucency, loss of disc height, loss of range of motion, or boney fusion.
  A Fusion patient was a considered to be a success if, and only if, ALL of the following criteria were met:
  Items numbered 1-3, above; 4. No re-operations required to modify the fusion site or correct a complication with an implant; and 5. Independent radiographic review confirmed strong evidence of fusion and no motion, visible gaps in fusion mass, loss of disc height, migration/subsidence, implant loosening, halos, or radiolucencies
Time Frame: 60 Months
Population: Patients who completed all 60 month visit analyses
Measure: Number; unit: percentage of overall successes
Arm/Group | 1-Level Fusion | 1-Level ProDisc | 1-Level ProDisc (Non-randomized) | 2-Level Fusion | 2-Level ProDisc | 2-Level ProDisc (Continued Access)
Number analyzed (Participants) | 52 | 134 | 39 | 57 | 116 | 0
percentage of overall successes | 50.0 | 53.7 | 56.4 | 50.9 | 55.2 |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at each visit through 60 month follow-up
Description: SYNCODE is a company defined medical coding category system for AEs
Arm/Group | 1-Level Fusion | 1-Level ProDisc | 1-Level ProDisc (Non-Randomized) | 2-Level Fusion | 2-Level ProDisc | 2-Level ProDisc (Continued Access)
Serious Adverse Events (participants affected / at risk) | 27/80 | 43/162 | 16/50 | 23/72 | 39/165 | 38/259
Other Adverse Events (participants affected / at risk) | 73/80 | 153/162 | 46/50 | 69/72 | 153/165 | 219/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Level Fusion (N=80) | 1-Level ProDisc (N=162) | 1-Level ProDisc (Non-Randomized) (N=50) | 2-Level Fusion (N=72) | 2-Level ProDisc (N=165) | 2-Level ProDisc (Continued Access) (N=259)
Additional Surgery Index Level (Surgical and medical procedures) | 8 (8) | 12 (12) | 2 (2) | 5 (6) | 2 (2) | 4 (4)
Blood Loss (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0 (0) | 2 (2) | 5 (5) | 4 (4)
Cardiovascular (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Death (General disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Infection (Infections and infestations) | 7 (7) | 6 (6) | 2 (2) | 5 (5) | 3 (3) | 2 (2)
Neurological (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Surgery - Adjacent Level (Surgical and medical procedures) | 2 (3) | 4 (6) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Surgery - Other (Surgical and medical procedures) | 12 (16) | 20 (24) | 7 (8) | 10 (12) | 19 (26) | 18 (23)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Level Fusion (N=80) | 1-Level ProDisc (N=162) | 1-Level ProDisc (Non-Randomized) (N=50) | 2-Level Fusion (N=72) | 2-Level ProDisc (N=165) | 2-Level ProDisc (Continued Access) (N=259)
Additional Surgery Index Level (Surgical and medical procedures) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 7 (7) | 0 (0) | 13 (17) | 10 (10) | 12 (12)
Burning or Dysesthetic Pain (General disorders) | 3 (3) | 8 (10) | 1 (1) | 2 (3) | 10 (10) | 10 (10)
Cardiovascular (Cardiac disorders) | 7 (9) | 10 (10) | 6 (6) | 6 (10) | 15 (18) | 14 (18)
Degenerative Disease Progression (General disorders) | 5 (6) | 17 (20) | 3 (3) | 1 (1) | 7 (7) | 3 (3)
Degenerative Disease Progression, Other Lumbar (General disorders) | 4 (4) | 11 (13) | 1 (1) | 7 (8) | 6 (7) | 7 (7)
Dermatological (Skin and subcutaneous tissue disorders) | 3 (4) | 8 (12) | 0 (0) | 6 (8) | 5 (8) | 9 (9)
Dermatological or Drug Allergy (Skin and subcutaneous tissue disorders) | 10 (12) | 22 (27) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Dizziness (General disorders) | 4 (4) | 4 (4) | 3 (3) | 4 (4) | 7 (7) | 8 (9)
Edema (Blood and lymphatic system disorders) | 5 (5) | 12 (17) | 1 (1) | 8 (8) | 12 (15) | 23 (27)
Fever (General disorders) | 10 (10) | 12 (13) | 2 (2) | 13 (15) | 31 (32) | 36 (36)
Gastrointestinal (Gastrointestinal disorders) | 25 (36) | 38 (54) | 15 (20) | 28 (49) | 66 (97) | 81 (127)
Genitourinary (General disorders) | 6 (6) | 19 (21) | 4 (4) | 9 (11) | 25 (28) | 31 (34)
Headache (General disorders) | 8 (8) | 12 (13) | 5 (5) | 10 (12) | 15 (19) | 24 (24)
Incision Site Related (Skin and subcutaneous tissue disorders) | 15 (16) | 10 (11) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 4 (4) | 5 (7) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Infection - Other non-wound related (Infections and infestations) | 4 (5) | 9 (11) | 4 (4) | 3 (3) | 11 (11) | 13 (13)
Infection - Superficial Wound with Incision Site Pain (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 6 (6) | 5 (5)
Infection, Not Index Level Related (Infections and infestations) | 6 (7) | 11 (14) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 5 (5) | 9 (11) | 3 (3) | 10 (12) | 22 (23) | 33 (33)
Migration Not Requiring Surgery (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Muscoloskeletal Spasms - Back (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 2 (2) | 9 (9) | 21 (24) | 27 (30)
Musculoskeletal Spasms - Leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 9 (10) | 7 (7)
Musculoskeletal Spasm (Musculoskeletal and connective tissue disorders) | 6 (7) | 13 (17) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neurological (Psychiatric disorders) | 11 (12) | 33 (46) | 7 (9) | 2 (2) | 4 (5) | 1 (1)
Non-Specific Musculoskeletal Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (9) | 0 (0) | 2 (2) | 8 (10) | 15 (16)
Numbness Peripheral Nerve or Non-Index Level Related (General disorders) | 9 (9) | 27 (35) | 6 (8) | 15 (20) | 30 (42) | 44 (56)
Other (General disorders) | 11 (15) | 20 (25) | 6 (8) | 13 (19) | 27 (36) | 23 (24)
Other Musculoskeletal (Musculoskeletal and connective tissue disorders) | 19 (26) | 26 (40) | 10 (12) | 11 (11) | 20 (24) | 30 (32)
Pain - Back (General disorders) | 34 (48) | 85 (129) | 23 (30) | 42 (55) | 67 (97) | 84 (107)
Pain - Back and Lower Extremities (General disorders) | 22 (25) | 44 (54) | 17 (23) | 23 (27) | 46 (63) | 43 (51)
Pain - Back and Lower Extremities with Numbness at Index Level (General disorders) | 5 (6) | 7 (8) | 1 (1) | 3 (3) | 8 (9) | 7 (7)
Pain - Back and Other (General disorders) | 7 (7) | 9 (9) | 3 (3) | 5 (5) | 15 (15) | 22 (23)
Pain - Incision Site (General disorders) | 6 (6) | 4 (4) | 0 (0) | 8 (9) | 19 (19) | 21 (21)
Pain - Lower Extremities (General disorders) | 20 (30) | 51 (75) | 17 (26) | 30 (43) | 61 (83) | 85 (110)
Pain - Lower Extremities with Numbness at Index Level (General disorders) | 2 (2) | 6 (8) | 2 (2) | 6 (9) | 8 (10) | 15 (16)
Pain Other (Not back, hip, leg) (General disorders) | 17 (20) | 46 (66) | 7 (10) | 16 (24) | 32 (38) | 37 (38)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 10 (10) | 2 (2) | 4 (5) | 10 (10) | 14 (14)
Pseudoarthrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Psychological (Psychiatric disorders) | 9 (11) | 25 (27) | 5 (6) | 12 (17) | 31 (38) | 32 (33)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (10) | 1 (1) | 8 (8) | 22 (23) | 21 (22)
Surgery - Index Level (Revision) (Surgical and medical procedures) | 4 (4) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 2 (2)
Surgery - Other (Surgical and medical procedures) | 5 (6) | 8 (9) | 4 (4) | 8 (9) | 34 (47) | 27 (28)
Vascular Injury (Blood and lymphatic system disorders) | 5 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel Damage/Bleeding, Minor (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Wound Issues - Other (General disorders) | 9 (9) | 7 (7) | 1 (2) | 6 (7) | 15 (17) | 23 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less